CLINICAL TRIAL: NCT06553820
Title: The Effect of MediYoga on Quality of Sleep, Blood Pressure and Quality of Life Among Older People: a Randomized Controlled Study
Brief Title: The Effect of MediYoga on Sleep Quality, Blood Pressure, and Quality of Life in Older Adults with Hypertension:
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Signe Stelling Risom, Associated Professor, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-24000021
Record Dates: First submitted 2024-08-08; First posted 2024-08-14 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Hypertension; Quality of Life; Quality of Sleep; Mental Health
Keywords: MediYoga; Hypertension; Mindfulness; Quality of life
MeSH Terms: conditions — Hypertension; Sleep Initiation and Maintenance Disorders; Psychological Well-Being | interventions — Yoga; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention group I, yoga 20 minutes x2 pr week (Experimental)
  Interventions: Behavioral: Intervention group I, Yoga 20 minutes x2 pr week
- Intervention Group II, yoga 40 minutes pr week (Experimental)
  Interventions: Behavioral: Intervention Group II, Yoga 40 minutes x2 pr week
- Control group, no intervention (Other): standard of care
  Interventions: Other: Control Group, No intervention

INTERVENTIONS:
Behavioral: Intervention group I, Yoga 20 minutes x2 pr week — App-based MediYoga exercises, 20 minutes per session, twice a week for a total of 10 weeks.
  Arms: Intervention group I, yoga 20 minutes x2 pr week
Behavioral: Intervention Group II, Yoga 40 minutes x2 pr week — App-based MediYoga exercises, 40 minutes per session, twice a week for a total of 10 weeks.
  Arms: Intervention Group II, yoga 40 minutes pr week
Other: Control Group, No intervention — standard of care only
  Arms: Control group, no intervention

SUMMARY:
The goal of this Randomized Controlled Trial is to test if an intervention consisting of Yoga can increase quality of sleep and health related quality of life and decrease BP. Secondary to explore and describe the implementation of a yoga intervention and the participants' experiences and perspectives on the intervention in a process evaluation.

The main question it aims to contribute knowledge about intervention of Yoga in a home environment for individuals with hypertension aged 65 years or older. Participants will (if they got selected into one of the two interventions groups), participate in Yoga exercises delivered by an app for 2 times a week for 10 weeks. Researchers will compare the intervention groups with the control group to see if Medi yoga has an effect in older people with hypertension.

DETAILED DESCRIPTION:
Hypertension is a common disease, and it is estimated that by 2025 one third of the world's population will have hypertension. The prevalence is increasing with age, and among older persons above the age of 90, 71% of women and 65 % of men have hypertension. Hypertension is related to cardiovascular illness, such as myocardial infarction, stroke, and death.

Poor subjective sleep quality has a significant association with an elevated risk of hypertension. Sleep disturbances are a significant risk factor for the development of depression in older adults. A recent review concluded that non-pharmacological interventions have the potential to improve self-reported sleep quality among older adults. There appears to be increasing evidence to support the long-term effect of virtual mindfulness-based interventions and their impact on sleep quality.

Several recent reviews have concluded that breathing exercises can be used as an alternative non-pharmacological therapy to lower blood pressure, but highlighted also that establish knowledge on duration and intensity needed to ensure the optimal effect.

The intervention follows the guidelines from MediYoga-MOSI, an evidence-based method developed in Sweden based on the classical kundalini tradition with elements from traditional Korean medicine and Ayurveda It has been adjusted to the Nordic context and is today used across the Swedish healthcare system.

The participants in the intervention group will participate in a breathing exercise, light yoga exercise and mindfulness intervention, as a review highlighted the effectiveness of combining these three elements. These programs will be translated into Danish and delivered via an app.

The participants will be randomly assigned to one of three groups: a control group, receiving usual care, or in one of two different intervention-groups in which the intervention takes place 2 times pr week for 10 weeks in addition to usual care. In group I the participants receive a 20-minute intervention, in group II the participants receive a 40-minute intervention. Participants receiving the intervention will be invited to participate online in follow-up sessions (after 2 and 6 weeks), where questions can be asked and adherence to intervention can be promoted

If the home-based MediYoga intervention proves effective, yoga exercises could serve as a supplementary treatment for blood pressure. Regular practice of MediYoga may also enhance patients' sleep quality and overall quality of life.

Statistical analysis will be performed using the Statistical Package for Social Sciences Program for the quantitative data. Descriptive statistics and inferential statistics will be used for data analysis. Descriptive statistics include frequency, percentage, mean and standard deviation, and inferential statistics include the chi-square test. The test of normality will be performed using the Shapiro-Wilk test. A paired t-test will apply to test for the significant differences within the groups and an unpaired t-test will be used to test for significant differences between the control and intervention groups. From comparable studies we expect an attrition rate of 50% since adherence to the intervention seem to be a challenge in comparable interventions where the patient must be physical active (like trials testing rehabilitation programs or yoga). Drop-out rate will be registered in a flowchart and both per protocol and intent-to-treat analyses will be performed. The level of significance was set as p<0.05. The analysis will be performed by a blinded statistician.

ELIGIBILITY:
Inclusion Criteria:

* Older people ≥65 years
* Diagnosed with hypertension.
* Speaking and reading Danish.
* Being able to consent.
* No comorbidity that restricts them from participating in the intervention.
* Being the owner or user of a smartphone or tablet.

Exclusion Criteria:

* Starting an antihypertension medication during the intervention
* Antihypertension medication is changed (more than 10% increase or reduction in an already used drug or a switch to another drug) during the intervention, which includes diuretics, ACE inhibitors, Calcium-blockers, or Angiotensin-2-blockers.
* Participated in mindfulness or yoga exercise regularly at any point during the last two years.
* Patients who have diagnosed sleep disorders for example sleep apnea or narcolepsy.
* Taking sleep medication regularly.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
sleep quality | 10 weeks
  Patient reported sleep quality measured on the PSQI (Pittsburg Sleep Quality Index). Minimum value: 0 Maximum value: 21 Higher scores: Indicate worse sleep quality The PSQI assesses sleep quality by compiling responses to questions covering various aspects of sleep, such as sleep duration, sleep problems, and daytime fatigue.
  A total score of 5 or higher generally indicates poor sleep quality.
  Between group change in baseline versus follow-up patient-reported sleep quality as assessed by the psqi questionnaire .

SECONDARY OUTCOMES:
Blood pressure | 10 weeks
  Reducing BP measured by self-monitoring in own home. Both Systolic blood pressure and diastolic blood pressure will be measured.
Health-related quality of life | 10 weeks
  improving health-related quality of life measured by SF-12 questionnaire. Minimum Value: 0 Maximum Value: 100 Higher Scores Mean: Better health-related quality of life
Mental health | 10 weeks
  with improving anxiety and depression, measured by the Hospital Anxiety and Depression Scale (HADS) Minimum Value: 0 Maximum Value: 21 (for each subscale: anxiety and depression; the total score can range from 0 to 42) Higher Scores Mean: Worse anxiety or depression. HADS assesses levels of anxiety and depression through separate subscales for each condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev and Gentofte Hospital, Herlev, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Risom SS, Amdi KV, Wahlstrom M, Rasmussen TB, Sharma S, Kabir ZN, Konradsen H. The effect of MediYoga on sleep-quality, blood pressure and quality of life among older people with hypertension: study protocol of a pragmatic randomized controlled trial. BMC Complement Med Ther. 2025 Mar 20;25(1):109. doi: 10.1186/s12906-025-04846-6. PMID 40114123